CLINICAL TRIAL: NCT02095002
Title: The Effect of Modified Valsalva Maneuver on Filling Degree of Internal Jugular Vein
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Geng guiqi, PhD, Fudan University
Other Study IDs: 2014315V
Record Dates: First submitted 2014-03-14; First posted 2014-03-24 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: the Filling of Jugular Vein Before Anesthesia With and Without Valsalva Maneuver
Keywords: modified valsalva maneuver, internal jugular vein

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

SUMMARY:
To explore the effect of modified valsalva maneuver on the filling degree of right internal jugular vein.

Method: The anteroposterior diameter and left-right diameter of right internal jugular vein in thirty adult gynecology patients were recorded during normal respiration and modified valsalva maneuver respectively.

Investigators hypothesis that modified valsalva maneuver would enchance the filling degree of right internal jugular vein.

ELIGIBILITY:
Inclusion Criteria:

- female patients age 18-60 years

Exclusion Criteria:

* heart or lung disease mental illness communication barriers.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: female genecology patients, age 18-60 years old; weight 45-70 kg; body mass index (BMI)>20 kg/m2 and <30 kg/m2; American Society of Anesthesiologists (ASA) grade I-II.
  The exclusion criteria were as follows: a history of chronic throat disease; upper respiratory tract infection within two weeks before surgery; and history of mental illness or communication barriers.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
the change of the diameter of right internal jugular vein after modified valsalva maneuver | up to 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Obstetrics & Gynecology Hospital, Fudan University, Shanghai, Shanghai Municipality, China